CLINICAL TRIAL: NCT05805553
Title: Role of Anabolic Steroid and Propranolol in Paediatric Burn- A Randomized Controlled Trial
Brief Title: Anabolic Steroid and Propranolol in Paediatric Burn
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Edward Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 126/RC/KEMU
Record Dates: First submitted 2021-01-26; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Arrest; Bone; Development; Growth
Keywords: Pediatric; Burn; Propranolol; Steroid; Growth; arrest
MeSH Terms: conditions — Heart Arrest; Burns | interventions — Propranolol; Nandrolone Decanoate

STUDY DESIGN:
Intervention Model Description: Three groups are made. one will receive steroid (control group). other will receive propranolol and third will receive both propranolol and steroid. their results will be compared
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): Propranolol will be given to this group
  Interventions: Drug: Propranolol
- group b (Experimental): steroid will be given
  Interventions: Drug: Nandrolone Decanoate
- group c (Experimental): both propranolol and steroids will be given
  Interventions: Drug: Propranolol; Drug: Nandrolone Decanoate

INTERVENTIONS:
Drug: Propranolol — 2mg/kg/day in 3-4 dividd doses
  Arms: Group A; group c
Drug: Nandrolone Decanoate — 1mg/kg weekly
  Arms: group b; group c

SUMMARY:
propranolol and anabolic steroids have a role in pediatric burn patients and their combined effects are to be studied here. They decrease the catabolic response to burn trauma and minimize the duration of growth arrest hence improving the outcome

DETAILED DESCRIPTION:
Burn is a major cause of morbidity and mortality worldwide; rate being seven times higher in low- and middle- income countries than high income countries. According to WHO, worldwide 11million people require medical attention secondary to burns. In Pakistan, 17% of burn patients have temporary disability while 18% suffer from a permanent disability Various studies have been done to improve patient outcome in terms of morbidity and mortality. Different medical interventions seem to have promising role in improving patient outcome in burn population.

Majority of pathological problems are due to catecholamines, an integral part of systemic metabolic drive, which increase approximately 10-fold as a response to injury . Hypermetabolic state has two aspects-the "ebb" and "flow" phases. The "ebb" phase lasts till first 48hours and has decreased metabolic rate and oxygen consumption while "flow" phase, which starts after resuscitation and has huge metabolic turnover, is the problematic one and needs intervention to decrease grave outcomes on patient's health. Systemic effects of catecholamines are significant once burned surface area increases more than 20% of the TBSA and persist for years . Various studies show that Propranolol and Oxandrolone have beneficial effects on decreasing morbidity and mortality in burn population Propranolol, a non-selective beta adrenergic blocker, has been used to minimize systemic effects of catecholamines and hypothetically results in anti-catabolic effects especially when given during ebb phase of the process i.e. decreases heart rate (HR) and blood pressure (BP) while during flow phase it increases hematocrit levels by increasing the renal erythropoietin secretion and decreases number of transfusions as well as blood loss during skin grafting "Herndon et al demonstrated that the cardiac effort was significantly reduced by 20% to 36% when the patients were given 2 mg/kg every 24 hours for 5 days. They determined that an ideal dose of 0.5 to 1.0 mg/kg intravenously every 6 to 8 hours should be given to adequately reduce left ventricular work without adversely affecting oxygen delivery or other cardiac functions" In another study done by Minifee et al, propranolol does not affect overall body delivery and consumption of oxygen but significantly decreases cardiac muscle requirement of oxygen . Moreover hyper-/hypo-glycemia, hypotension, azotemia, hypothermia, arrythmias and peripheral ischemia are also not observed as adverse effects . Another study by Baron et al showed that prolonged administration of oral or IV propranolol does not have an adverse effect on morbidity or mortality

Anabolic steroid (Oxandrolone/nandrolone) has a definite role in building up body's protein stores. Unlike testosterone, its adverse effects, acne, hirsutism, behavioral changes and liver functions are not documented, so they are considered safe. Use of oxandrolone alone and in combination with propranolol has a definitive effect as anti-catabolic agent and helps in better recovery and long-term outcomes on child's growth and decreases cardiac load.

A study done by Sylvia Ojeda et al at university of Texan in 2018 showed that propranolol is both safe and effective in managing the cardiovascular effects of hypermetabolic state in burn patients. A couple of other studies show that both propranolol and oxandrolone have a role in reducing the burden of disease in burn but data is lacking on effects of administration of both the drugs combined. Moreover, how the medication will affect our population is yet to be determined. This study will help us compare the effects of both drugs in our population and decrease the morbidity and mortality in burn patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting within 48 hours of burn
* more than 20% and less than 40 %of TBSA burn (measured via modified rule of nine for pediatric burn according to age)
* age 2-12 years (as safety of anabolic steroids is not established in <2years of age)
* Scald and flame burn

Exclusion Criteria:

* Diabetics (diagnosed before hospital admission)
* Renal disease (diagnosed before hospital admission)
* Asthmatics (on medication previously)
* Cardiac anomalies (previously diagnosed)
* Patients requiring cardiac support (norepinephrine, dobutamine at any dose and dopamine >7ug/kg).
* All 4 limbs burnt

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 114 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-09-28 (Estimated); Study Completion 2023-09-28 (Estimated)

PRIMARY OUTCOMES:
reversal of growth arrest | at 1 year after burn
  BMI in kg/m^2
Bone mineral density measure | at 1 year
  Bone mineral density as g/cm^2 (Z-score)

SECONDARY OUTCOMES:
no of blood transfusions | at 60 days
  number of blood transfusions during hospital stay

CONTACTS AND LOCATIONS:
Locations (1):
- King Edward Medical University, Mayo Hospital, Lahore, Punjab Province, Pakistan